CLINICAL TRIAL: NCT05676996
Title: Investigation of the Effect of Attachment-Based Support Given in the Perinatal Period on Prenatal Bonding, Early Mother-Infant Bonding Indicators and Maternal Bonding
Brief Title: Investigation of the Effect of Attachment-Based Support Given in the Perinatal Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Özge Karakaya Suzan, Principal Investigator, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Attachment-Based Support
Record Dates: First submitted 2022-12-30; First posted 2023-01-09 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Attachment Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- attachment-based support group (Experimental): In addition to the routine follow-ups and trainings that the pregnant women in the intervention group can receive from the hospital, they will be included in the "Attachment Based Support Program". Within the scope of the 1st stage of this support; A mobile application. There are 12 videos on connecting in the mobile application. These videos were shot by the researcher in a professional studio. 22nd-26th of pregnancy. The participants included in the study during the weeks of participation installed this mobile application on their phones during participation. It was requested to complete watching the videos by 36 weeks. In the second phase of Attachment-Based Support, breastfeeding and skin-to-skin contact support are provided to mothers on postpartum day 0.
  Interventions: Other: attachment-based support
- routine follow-up control group (No Intervention): The control group pregnants were left to the routine follow-up of the hospitals during their pregnancy and postpartum period. In this follow-up; When pregnant women apply to the outpatient clinic services of the hospital, appointments are made for their monthly routine follow-up. Information and practices that support mother-infant attachment in attachment-based support modules are not included in these trainings.

INTERVENTIONS:
Other: attachment-based support — attachment-based support application; It includes video-based trainings on attachment via mobile application and breastfeeding and skin-to-skin contact support for mothers on postpartum day 0.
  Arms: attachment-based support group

SUMMARY:
It is important that effective intervention programs are developed and implemented in our country by identifying risk factors in the early period. In this aspect, the work is unique. Unlike the studies in the literature, it is a unique study in terms of determining the risky population that needs to be questioned and strengthened during the prenatal attachment of expectant mothers during pregnancy, and creating a program where mothers can receive uninterrupted support for 24 hours.

DETAILED DESCRIPTION:
Mother-infant attachment is also an important factor for adaptation to the maternal role. Attachment begins in the prenatal period and continues in the postnatal period. Attachment in the prenatal and postnatal period is related to each other . Abasi et al. (2013) stated that the attachment strengthening intervention program applied to pregnant women can positively affect maternal mental health, fetal health and ultimately child health. In the study of Akbarzadeh et al. (2016), investigators found that by educating mothers on attachment skills, the bond between mothers and fetuses is strengthened and the mental health of babies can be improved after birth. It has been reported that prenatal attachment affects postnatal parenting roles and plays an important role in the child's growth and development. Therefore, mother-infant attachment begins in the prenatal period, not in the neonatal period. Peppers and Knapp in their study; investigators found that the mother's contact with her stillborn baby did not affect the mother's grief process and suggested that mother-infant attachment begins in the prenatal period, not in the newborn period. Prenatal attachment can be affected by many factors. In the studies carried out; It has been observed that education level, desired pregnancy status, gestational week, feeling fetal movements, coping styles with stress and anxiety experienced during pregnancy, body image perceptions, emotional intelligence and social support perceptions of pregnant women, and the support given to the mother before birth affect prenatal attachment. For this reason, it is important to determine prenatal attachment behaviors during pregnancy, to examine the factors affecting attachment behaviors, to identify pregnant women with low attachment levels, as they may have positive contributions to mother-infant health in the prenatal and postnatal period. When investigators examine the international literature, although there are studies to support attachment, there is a study in our country for the population that can be strengthened by determining the prenatal attachment level. It is important that effective intervention programs are developed and implemented in our country by identifying risk factors in the early period. In this aspect, the work is unique. Unlike the studies in the literature, it is a unique study in terms of determining the risky population that needs to be questioned and strengthened during the prenatal attachment of expectant mothers during pregnancy, and creating a program where mothers can receive uninterrupted support for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

be 19 years or older 21 and 26. Primigravida at gestational week Having had a normal delivery Watching all the videos within the scope of Attachment-Based Support Program by the pregnant women in the intervention group Being literate Pregnancy with only one baby The baby is at term Being the mother of the primary caregiver Volunteering to participate in the research The absence of any health problems of the mother and the baby Absence of a physician-diagnosed psychiatric disease in the mother Having a smart phone and wireless internet Pregnant women who answered "No" to Question 34 on the Pregnant Introductory Information Form and did not get a full score from the "Maternal Antenatal Attachment Scale"

Exclusion Criteria:

* The development of a situation that prevents the mother from participating in education during pregnancy
* Unwillingness to continue working
* A situation that prevents the mother and baby from staying in the same room in the postpartum period
* Severe trauma or loss of the mother during pregnancy

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Enrollment: 70 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Prenatal attachment of pregnant women who participated in the attachment-based support program in the perinatal period compared to those who did not participate is higher. | 22.-26. pre-test between weeks
  prenatal attachment scale; There are a total of 19 items in the scale, which focuses on the pregnant woman's feelings, attitudes and behaviors towards the fetus. The scale is in a 5-point Likert type and each item is scored between 1 and 5 (5=represents very strong feelings towards the fetus; 1=represents the absence of feelings towards the fetus). A high score from the scale indicates a high degree of attachment.
Pregnant women who participated in the Attachment-Based Support Program during the perinatal period showed more early mother-infant attachment symptoms than those who did not. | this scale will be administered to mothers on postpartum day 0.
  The scale of early mother-infant attachment indicators is an observational scale consisting of 13 items. The lowest 0 and the highest 26 points are taken from the scale. As the scores obtained from the scale increase, attachment increases.
Pregnant women who participated in Attachment-Based Support Program in the perinatal period had higher maternal attachment than those who did not. | postpartum 1st month
  The maternal attachment scale is a scale applied at the earliest postpartum 1st month. The lowest score to be obtained from the scale varies between 26 and the highest score between 104. A high score from the scale indicates a high level of maternal attachment.
Prenatal attachment of pregnant women who participated in the attachment-based support program in the perinatal period compared to those who did not participate is higher. | post-test at 36 weeks
  prenatal attachment scale; There are a total of 19 items in the scale, which focuses on the pregnant woman's feelings, attitudes and behaviors towards the fetus. The scale is in a 5-point Likert type and each item is scored between 1 and 5 (5=represents very strong feelings towards the fetus; 1=represents the absence of feelings towards the fetus). A high score from the scale indicates a high degree of attachment.

CONTACTS AND LOCATIONS:
Overall Officials: Nursan CİNAR, PhD, Study Director — Sakarya University
Locations (1):
- Sakarya University Training and Research Hospital, Adapazarı, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
can be published after the work is completed.